CLINICAL TRIAL: NCT05654480
Title: Combating Diagnostic Wandering and Impasse for Cystic Fibrosis: Assessment of Patients Not Concluded After Neonatal Screening of Cystic Fibrosis
Brief Title: Combating Diagnostic Wandering and Impasse for Cystic Fibrosis
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Societe Francaise de la Mucoviscidose (Other)
Collaborators: Vaincre la Mucoviscidose (Other)
Responsible Party: Principal Investigator, Isabelle SERMET-GAUDELUS, Professor, Societe Francaise de la Mucoviscidose
Other Study IDs: CF impasse
Record Dates: First submitted 2022-11-25; First posted 2022-12-16 (Actual); Last update posted 2022-12-16 (Actual); Status verified 2022-12

CONDITIONS: Cystic Fibrosis
MeSH Terms: conditions — Cystic Fibrosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
After cystic fibrosis (CF) neonatal screening, some children remain with a not concluded diagnosis. In France, the medical follow-up is not standardized, some of them may be lost of follow-up. The aim of the study is to identify children at risk of developing CF. Other children carry mutation at risk of CFTR related disorder (CFTR-RD) but remain asymptomatic during childhood. The aim of the study is to evaluate those children by microbiology, respiratory function test and lung imaging tests to reclassify them in the CFTR spectrum.

DETAILED DESCRIPTION:
Cystic fibrosis (CF) is a life-limiting genetic disorder related to the mutation of the CF Transmembrane Conductance Regulator (CFTR) gene. Cystic fibrosis neonatal screening in France has been generalized in 2002. Patients with hypertrypsinemia and two CF mutations are diagnosed CF and followed in CF center with standards of care.

But some children with hypertrypsinemia may have an intermediate chloride sweat test and only one CFTR mutation, or a negative sweat test and two CFTR mutations at least one of which is of unknown pathogenicity.

Some other patients may present with two CFTR-RD mutations and may unravel a monosymptomatic disease in adulthood (CFTR-related disorder) such as congenital bilateral absence of vas deferens (CBAVD), acute recurrent or chronic pancreatitis, disseminated bronchiectasis, chronic rhinosinusitis...We have very few data about age of onset, type of symptoms, and infraclinical disease.

Patients will be identified according to neonatal screening data and genetic database, and will undergo clinical evaluation, pancreatic and lung disease evaluation to reclassify them in the CFTR spectrum.

ELIGIBILITY:
Inclusion Criteria:

* undiagnosed patients with hypertrypsinemia at CF neonatal screening and :

  1. either an intermediate chloride sweat test (30-59 mmol/L) and at most one CFTR mutation
  2. or negative chloride sweat test (< 30 mmol/L) and two CFTR mutations one of wich is of unknown significance (VUS)
* patients with two CFTR mutations at least one of which is of Varying Clinical Consequence according to "CFTR2" database or "CFTR-RD" according to "CFTR-France" database.

Exclusion Criteria:

* CF patients with 2 CF causing mutations

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Adult patients and pediatric patients evaluated at neonatal screening and :
  1) either an intermediate chloride sweat test (30-59 mmol/L) and at most one CFTR mutation (2) or negative chloride sweat test (< 30 mmol/L) and two CFTR mutations one of wich is of unknown significance (VUS)
  Adult and pediatric patients carrying at least two CFTR mutations one of which at least is of Varying Clinical Consequence according to "CFTR2" database or "CFTR-RD" according to "CFTR-France" database.
Sampling Method: Non-Probability Sample
Enrollment: 400 (Estimated)
Dates: Start 2023-01-02 (Estimated); Primary Completion 2024-05-01 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
sputum bacteriology | previous and at inclusion
  bacteria, fungi and mycobacteria

SECONDARY OUTCOMES:
spirometry | previous and at inclusion
  Forced Expiratory Volume in 1 second, Forced VItal capacity
Lung Clearance index (LCI) | previous and at inclusion
  Lung Clearance Index 2.5 %
Plethysmography | previous and at inclusion
  Residual volume
lung imaging | previous and at inclusion
  Low dose CT scan
sweat test | previous and at inclusion
  chloride sweat concentration
pulmonary exacerbations | previous to inclusion
  number of pulmonary exacerbations
pancreatic function | previous and at inclusion
  fecal elastase
liver function | previous and at inclusion
  liver function test
liver ultrasound | previous and at inclusion
  liver parenchyma evaluation

CONTACTS AND LOCATIONS:
Overall Officials: Christophe Marguet, MD, Study Director — Societe Francaise de la Mucoviscidose
Locations (1):
- Necker Hospital, Paris, France